CLINICAL TRIAL: NCT06429891
Title: Research on Early Diagnosis and Clinical Transformation of Nuclide Probe Based on Bioorthogonal-gastric Cancer Mucin Target Visualization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hua Zhu (Other)
Responsible Party: Sponsor-Investigator, Hua Zhu, Principal Investigator, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024KT68
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-16A (Experimental): All study participants will be allocated to this arm (single-arm study). Study participants will undergo 89Zr-16A PET/CT scans.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — All study participants will undergo one 18F-FDG PET/CT scan.

SUMMARY:
The symptoms of early gastric cancer are extremely insidious and most patients are identified as advanced at the time of initial diagnosis. Starting from the clinical needs, this project selects solid tumors and pathogenic glycoprotein synthesis of key glycopeptide antigen determinant mucin (MUC) family of multiple molecules as the research object. Based on the digestive system tumor research cohort established in the early stage, this project intends to verify the tumor microenvironment characteristics of the MUC family and gastric cancer treatment resistance through immunohistochemistry, COSMC gene sequencing and other technologies, and screen key MUC family proteins. Based on the discovery of differential recognition of COSMC deficient cells by antibodies, MUC1-targeted specific monoclonal antibody was developed. Further development of spatial mucinomics based on laser ablation inductively coupled plasma mass spectrometry (LA-IPC-MS) and spatial metabolome based on desorption electrospray mass spectrometry (DESI-MS) to analyze the structure and immunosuppressive mechanism of key gastric cancer glycoprotein MUC. After obtaining key targeted antibodies, with the help of biological orthogonal and click chemistry technology, the original clinical translational research based on mucin targeting was carried out, and a high-affinity nuclide conjugate drug (RDC) with "triple binding" of gastric cancer mucin was constructed and clinical translational research was carried out, which provided new ideas for the accurate diagnosis and treatment of gastric cancer in the early stage.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years old; ECOG 0 or 1;
2. Patients with solid tumor confirmed by histopathology;
3. Patients with imaging confirmed measurable lesions;
4. life expectancy >=12 weeks.

Exclusion Criteria:

1. Significant hepatic or renal dysfunction;
2. ls pregnant or ready to pregnant;
3. Cannot keep their states for half an hour;
4. Refusal to join the clinical study;
5. Suffering from claustrophobia or other mental diseases；
6. Any other situation that researchers think it is not suitable to participate in the experiment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 2 years
  The uptake of the tracer (89Zr-16A) in solid tumor lesions or suspected tumor lesions by measuring SUV on PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhu, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China